CLINICAL TRIAL: NCT01113879
Title: Exercise as an Adjuvant to Aphasia Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C7175-M
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Aphasia
Keywords: rehabilitation; aphasia; exercise; BDNF
MeSH Terms: conditions — Aphasia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study used a single-subject, multiple-baseline design across behaviors. Following assessment and baseline procedures, participants completed 2 therapy periods: Block 1 was aphasia therapy alone, and Block 2 was aphasia therapy plus aerobic exercise or stretching.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aphasia therapy with an exercise adjuvant (Experimental): Aphasia therapy for anomia: The treatment is a traditional lexical/semantic stimulation approach during which subjects will attempt to name drawings of objects.
  Aerobic exercise: An aerobic exercise intervention will target cardiorespiratory fitness by progressing from 50-70% of the participants' maximum heart rate.
  Interventions: Behavioral: Aerobic exercise
- Aphasia therapy with a stretching adjuvant (Placebo Comparator): Aphasia therapy for anomia: The treatment is a traditional lexical/semantic stimulation approach during which subjects will attempt to name drawings of objects.
  Stretching: Stretching will occur for 50 minutes a day, three days/week for 12 weeks.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Aerobic exercise — An aerobic exercise intervention will target cardiorespiratory fitness by progressing from 50-70% of the participants' maximum heart rate.
  Arms: Aphasia therapy with an exercise adjuvant
Behavioral: Stretching — Stretching will occur for 50 minutes a day, three days/week for 12 weeks.
  Arms: Aphasia therapy with a stretching adjuvant

SUMMARY:
The purpose of the study is to reveal if individuals who participate in aerobic activity demonstrate greater improvement in language abilities than patients who do not participate in aerobic activity.

DETAILED DESCRIPTION:
The objective of this research project is to reveal if individuals who participate in aerobic activity demonstrate greater improvement in language abilities with treatment than patients who do not participate in aerobic activity. As secondary objectives, we will determine if there is a direct relationship between either brain efficiency or increases in Brain Derived Neurotrophic Factor (BDNF) after exercise and higher learning rates in aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke aphasia
* at least 6 months post-stroke
* at least minimally intact auditory verbal comprehension
* pre-morbidly right handed
* native English speaker

Exclusion Criteria:

* contraindications for fMRI (metal implants, claustrophobia)
* inability to pass an exercise tolerance test
* significant depression
* uncorrected hearing or vision problems
* severe apraxia of speech
* regularly perform 20 minutes of cardiovascular exercise 3 times per week

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy M. Harnish, PhD CCC/SLP, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Brooks Rehabilitation Clinical Research Center, Jacksonville, Florida

REFERENCES:
- [Derived] Harnish SM, Rodriguez AD, Blackett DS, Gregory C, Seeds L, Boatright JH, Crosson B. Aerobic Exercise as an Adjuvant to Aphasia Therapy: Theory, Preliminary Findings, and Future Directions. Clin Ther. 2018 Jan;40(1):35-48.e6. doi: 10.1016/j.clinthera.2017.12.002. Epub 2017 Dec 23. PMID 29277374
- See also: Click here for more information about this study: Exercise as an Adjuvant to Aphasia Therapy — http://www.brrc.research.va.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Aphasia Therapy Alone, Then With Exercise: Aphasia therapy for anomia: The treatment is a traditional lexical/semantic stimulation approach during which subjects will attempt to name drawings of objects.
  Aerobic exercise: An aerobic exercise intervention will target cardiorespiratory fitness by progressing from 50-70% of the participants' maximum heart rate.
  Following assessment and baseline procedures, participants completed 2 therapy periods: Block 1 was aphasia therapy alone, and Block 2 was aphasia therapy plus an aerobic exercise or stretching adjuvant.
- Aphasia Therapy Alone, Then With Stretching: Aphasia therapy for anomia: The treatment is a traditional lexical/semantic stimulation approach during which subjects will attempt to name drawings of objects.
  Stretching: Stretching will occur for 50 minutes a day, three days/week for 12 weeks.
Period: Period 1: Block 1
Arm/Group | Aphasia Therapy Alone, Then With Exercise | Aphasia Therapy Alone, Then With Stretching
Started | 7 | 2
Completed | 5 | 2
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Period 2: Block 2
Arm/Group | Aphasia Therapy Alone, Then With Exercise | Aphasia Therapy Alone, Then With Stretching
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aphasia Therapy With an Exercise Adjuvant | Aphasia Therapy With a Stretching Adjuvant | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (12.5) | 44.5 (10.6) | 57.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 2 | 9
Boston Naming Test [Mean (Full Range); unit: units on a scale] — The Boston Naming Test measures picture naming abilities. The range is 0-60 with higher scores corresponding with better naming abilities.
  units on a scale | 20.6 [10 to 43] | 21.5 [4 to 39] | 20.9 [4 to 43]
Western Aphasia Battery [Mean (Full Range); unit: units on a scale] — The Western Aphasia Battery Aphasia Quotient range is 0-100 with higher scores demonstrating better language abilities. A score of less than 93.8 is the clinical cutoff for the diagnosis of aphasia.
  units on a scale | 58.6 [43.5 to 80.7] | 60.1 [35.8 to 84.4] | 59 [35.8 to 80.7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Picture Naming Abilities as Measured by Tau U Effect Size Weighted Means
Description: Tau-U effect sizes of <0.20 were considered small; 0.20 to <0.60 moderate; 0.60 to <0.80 large, and >=0.80 very large. Weighted Tau-U averages in exercise participants and stretching participants were calculated in each block using an online web-based calculator (http://www.singleresearch.org/calculators/tau-u). In the present analysis, any baseline trends over 0.10 were adjusted.
Time Frame: administered before and after each of two, two week aphasia therapy blocks
Measure: Mean (80% Confidence Interval); unit: Tau U effect size weighted mean
Arm/Group | Aphasia Therapy With an Exercise Adjuvant | Aphasia Therapy With a Stretching Adjuvant
Number analyzed (Participants) | 5 | 2
Tau U effect size weighted mean
  Weighted Tau U for Block 1 | 0.83 [0.67 to 1.00] | 0.75 [0.49 to 1.00]
  Weighted Tau U for Block 2 | 0.88 [0.71 to 1.00] | 0.77 [0.50 to 1.00]
Statistical Analysis 1: Comparison: Aphasia Therapy With an Exercise Adjuvant; Weighted Tau U effect size mean values in Block 1 of treatment (no aerobic exercise or stretching) were compared to weighted Tau U mean values in Block 2 of treatment (aerobic exercise or stretching adjuvant); Test type: Other; p < 0.001, Weighted Tau U

2. Secondary Outcome: Change in Serum Brain-derived Neurotrophic Factor (BDNF) Levels With Exercise
Description: The baseline BDNF levels in participants (ie, the 2 measures prior to the exercise or stretching interventions) showed a great deal of intraparticipant variation. Hence, in an attempt to minimize the intraparticipant variability, we calculated the mean values from samples 1 and 2 to obtain a baseline BDNF measure, samples 3 and 4 to obtain a BDNF measure in the first 6 weeks of aerobic exercise or stretching, and samples 5 and 6 to obtain a measure in the last 6 weeks of the exercise or stretching intervention.
Time Frame: six samples collected over a 16 week period
Population: Complete BDNF datasets from 5 of the 7 participants who completed the study were available. BDNF data from the remaining two participants were not collected due to the PI and study team moving locations and no longer having access to the facilities.
Measure: Number; unit: participants
Arm/Group | Aphasia Therapy With an Exercise Adjuvant | Aphasia Therapy With a Stretching Adjuvant
Number analyzed (Participants) | 4 | 1
participants
  BDNF increased from baseline to six weeks adjuvant | 0 | 1
  BDNF increased from first 6 weeks to last 6 weeks | 4 | 0
  BDNF decreased from baseline to six week adjuvant | 4 | 0
  BDNF decreased from first 6 weeks to last 6 weeks | 0 | 1

ADVERSE EVENTS:
Arm/Group | Aphasia Therapy With an Exercise Adjuvant | Aphasia Therapy With a Stretching Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No